CLINICAL TRIAL: NCT06514417
Title: Efficacy of Ultrasound - Guided External Oblique Intercostal Plane Block for Patients Undergoing Upper Abdominal Surgeries: A Randomized Controlled Trial
Brief Title: External Oblique Intercostal Plane Block for Patients Undergoing Upper Abdominal Surgeries
Acronym: EOINB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Ayman Ahmed Rady (Unknown); Ahmed Mohamed Helwa (Unknown)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7/2023ANET12
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external oblique intercostal block (Active Comparator): receive US-guided external oblique intercostal block after induction
  Interventions: Other: US-guided external oblique intercostal block
- No block (No Intervention): receive postoperative morphine on patient request

INTERVENTIONS:
Other: US-guided external oblique intercostal block — After induction of general anesthesia, external oblique intercostal block will be performed (8) under ultrasonographic guidance with transportable ultrasound device ( Sonosite ,superficial probe ,14-15 MHz).
  the patient will be positioned supine, and a linear ultrasound transducer will be placed in the sagittal plane between the midclavicular and anterior axillary lines at the level of sixth rib. 20 ml of bupivacaine 0.25% will be injected between the plane of the external oblique and the intercostal muscles. The drug will be injected after a negative aspiration.
  The contralateral side block will be performed in a same manner.
  Arms: external oblique intercostal block

SUMMARY:
Ithe study will evaluate the analgesic efficacy of external oblique intercostal block for patients undergoing upper abdominal surgeries

DETAILED DESCRIPTION:
Patients will be randomly divided into two equal groups using SPSS. Group A: will receive US-guided external oblique intercostal block after induction Group B: will receive postoperative morphine on patient request. Study design: prospective controlled randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Selected patients will be more than 21 years old with ASA physical status I & II scheduled for upper abdominal surgeries

Exclusion Criteria:

Uncooperative patients.

* Patients who have allergy to any of the used drugs.
* Patients who are on opioids.
* Known abuse of alcohol or medication.
* Local infection at the site of injection or systemic infection.
* Pregnancy
* Patients with coagulation disorders or on anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale . | 24 hours
  postoperative pain that evaluated by visual analogue pain scale(a scale from 0 to 10 where 0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain)

SECONDARY OUTCOMES:
total perioperative analgesics requirements | 24 hours
  Milligram

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No